CLINICAL TRIAL: NCT05097339
Title: cArdiopulmonary exerCise Test Assessing Multiple bIOmarkers iN Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Indigo Diabetes NV (Industry); Université Montpellier (Other); Campus Bio-Medico University (Other); University of Padova (Other)
Responsible Party: Principal Investigator, Christophe De Block, Prof Dr Christophe De Block, Head of the Department of Endocrinology, Diabetology and Metabolism, Principal Investigator, Clinical Professor, University Hospital, Antwerp
Other Study IDs: ACTION1
Record Dates: First submitted 2021-09-22; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: exercise; biomarker; glucose; lactate; ketones; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Ketosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — Venous blood samples were analysed for glucose, lactate and ketone values with YSI technology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with type 1 diabetes: Patients with type 1 diabetes perform a morning Symptom Limited Maximal Exercise Test (CPET) or a 60-minute morning Aerobic Test (AEX) at 60% VO2peak

SUMMARY:
Collection of venous blood samples in male T1D patients to evaluate the behavior of different biomarkers (beta-hydroxybutyrate, lactate, glucose) during and after morning Aerobic (60% of VO2 max) and Symptom Limited Maximal Exercise Test.

DETAILED DESCRIPTION:
Compare values and trends of different biomarkers (glucose, lactate and beta-hydroxybutyrate) before, during and after morning aerobic and symptom limited maximal exercise (cycling) to predict glycemic fluctuations (hypo- and hyperglycemic events) during and after exercise in order to create treatment algorithms to prevent these events.

Endpoint:

• Evaluate values and trends of glucose, lactate and beta-hydroxybutyrate before, during and after morning exercise in venous blood.

ELIGIBILITY:
Inclusion Criteria:

* Male adults (18-40 years old) with T1D, diagnosed since > 1 year
* Using a CGM (Dexcom G5) or willing to wear a CGM (Dexcom G5) for the duration of the study.

The CGM must be applied >48h before the exercise test

* Participants are on intensified insulin therapy (MDI) or insulin pump therapy (CSII)
* 6% ≤ HbA1c ≤ 8%
* Having a self-reported moderate activity level on the iPAQ (Internationally Physical Activity Questionnaire).
* C-peptide <0.2 nmol/l
* The Physical Activity Coefficient has not changed in the 2 months prior to the first Exercise Test.
* 20kg/m2 < BMI < 25kg/m2

Exclusion Criteria:

* Recently diagnosed T1D (< 12mo)
* Participants not on MDI or CSII
* Musculoskeletal disorder that affects cycling or is a contra-indication for vigorous physical activity
* Cardiorespiratory disease or ECG abnormality that is a contra-indication for vigorous physical activity
* Having an acute illness (e.g. influenza) that interferes with glucose metabolism
* Having a metabolic disorder (different from diabetes) or takes drugs known to have significant interference with glucose metabolism, such as systemic corticoids as judged by the investigator
* Current treatment with drugs known to have significant interference with glucose metabolism, such as systemic corticoids as judged by the investigator
* Presence of concomitant pathology such as heart failure, liver failure, kidney failure defined as eGFR <45mL/min
* Patient not able or willing to sign the patient informed consent

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult male participants, aged 18-40 years, with Type 1 Diabetes (T1D) treated with Multiple Daily Insulin injections (MDI) and Continuous Subcutaneous Insulin Injections (CSII)
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Change in glucose concentration during and after morning Aerobic and Symptom Limited Maximal Exercise Test | Blood sampling was done before the exercise, every 3 minutes for CPET and every 5 minutes for AEX during the exercise and every 15 minutes during the first hour of recovery and every 20 minutes during the rest of the 6-hour follow-up.
  Glucose levels in mg/dL during and after morning Aerobic (60 minutes at 60% of VO2 max) and Symptom Limited Maximal Exercise Test (AEX & CPET), measured in 21 patients through YSI (YSI Life Sciences, Yellow Springs, OH)
Change in lactate concentration during and after morning Aerobic and Symptom Limited Maximal Exercise Test | Blood sampling was done before the exercise, every 3 minutes for CPET and every 5 minutes for AEX during the exercise and every 15 minutes during the first hour of recovery and every 20 minutes during the rest of the 6-hour follow-up.
  Lactate levels in mmol/mol during and after morning Aerobic (60 minutes at 60% of VO2 max) and Symptom Limited Maximal Exercise Test (AEX & CPET), measured in 21 patients through YSI (YSI Life Sciences, Yellow Springs, OH)
Change in ketone concentration during and after morning Aerobic and Symptom Limited Maximal Exercise Test | Blood sampling was done before the exercise, every 3 minutes for CPET and every 5 minutes for AEX during the exercise and every 15 minutes during the first hour of recovery and every 20 minutes during the rest of the 6-hour follow-up.
  Ketone levels (Beta-hydroxybutyrate) in mmol/mol during and after morning Aerobic (60 minutes at 60% of VO2 max) and Symptom Limited Maximal Exercise Test (AEX & CPET), measured in 21 patients through YSI (YSI Life Sciences, Yellow Springs, OH)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe De Block, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Ridder F, Ledeganck KJ, De Winter B, Braspenning R, Delbeke D, Renard E, Pozzilli P, Pieralice S, Vissers D, De Block C. Trends of glucose, lactate and ketones during anaerobic and aerobic exercise in subjects with type 1 diabetes: The ACTION-1 study. Diabetes Metab Res Rev. 2022 Sep;38(6):e3537. doi: 10.1002/dmrr.3537. Epub 2022 May 21. PMID 35533265